CLINICAL TRIAL: NCT06029205
Title: The Effect of Conscious Awareness-Based Educatıon on Perceived Work Stress in Nurses
Brief Title: Mindfulness Training in Nurses and Its Effect on Work Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Merve ATAÇ ÖKSÜZ, lecturer doctor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: merveatac
Record Dates: First submitted 2023-07-11; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Nursing Caries; Consciousness, Level Altered
Keywords: nurse; work stress; awareness
MeSH Terms: conditions — Consciousness Disorders; Occupational Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Conscious Awareness-Based Educatıon on Perceived Work Stress in Nurses (Experimental): mindfulness-based education
  Interventions: Behavioral: Conscious Awareness-Based Educatıon
- The effect of stress coping training on nurses (Placebo Comparator): stress coping training
  Interventions: Behavioral: Stress coping training

INTERVENTIONS:
Behavioral: Conscious Awareness-Based Educatıon — The effect of Conscious Awareness-Based Education on nurses
  Arms: The Effect of Conscious Awareness-Based Educatıon on Perceived Work Stress in Nurses
Behavioral: Stress coping training — The effect of stress coping training on nurses
  Arms: The effect of stress coping training on nurses

SUMMARY:
The aim of the study, which was planned in the experimental design type, was to determine the effect of the mindfulness-based stress reduction training on nurses' job stress. The sample of the study consisted of 70 nurses (35 in the experimental group, 35 in the control group) working in a university hospital in Çanakkale. The mindfulness-based stress reduction training was carried out as a group, once a week, for 8 weeks in total.

DETAILED DESCRIPTION:
One of the most important problems of nurses in Turkey is the stress they experience at work. This stress experienced in the workplace is accompanied by consequences such as depression, anxiety, and decreased job satisfaction. Therefore, it is clear that addressing the stress associated with the nursing profession is an urgent problem. The aim of the study, which was planned in the experimental design type, was to determine the effect of the mindfulness-based stress reduction training on nurses' job stress. The sample of the study consisted of 70 nurses (35 in the experimental group, 35 in the control group) working in a university hospital in Çanakkale. The mindfulness-based stress reduction training was carried out as a group, once a week, for 8 weeks in total. The Personal Information Form, the Job Stress Scale, the Mindful Attention Awareness Scale, and the Rosenbaum's Learned Resourcefulness Scale were used for data collection. A total of three follow-ups were conducted to the nurses before the training, at the end of the training, and 3 months after the training. Descriptive analysis, Chi-square test, Independent Samples T-test, Dependent Samples T-test, and one-way analysis of variance were used in the analysis of the research data.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in the relevant health practice and research hospital
* Not having participated in any mindfulness-based training program before

Exclusion Criteria:

* Working as an executive nurse
* Not attending any session of the 8-week training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
The Effect of Conscious Awareness-Based Educatıon on Perceived Work Stress in Nurses | 8 week
  the Job Stress Scale (The maximum score that can be taken from the scale is 50, the minimum score is 10, and less than 12 points indicates a low-stress situation, between 12-30 points a stressful situation, and above 30 points a high-stress situation)
The Effect of Conscious Awareness-Based Education on Awareness in Nurses | 8 week
  the Mindful Attention Awareness Scale (The total score that can be obtained from thescale ranges from 0 to 90)
Learned Resourcefulness Effect of Conscious Awareness-Based Education on Nurses | 8 week
  Rosenbaum's Learned Resourcefulness Scale (A score between a minimum of 36 and a maximum of 180 can be obtained from the scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart Universty Hospital, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No